CLINICAL TRIAL: NCT00621140
Title: A Randomised, Double-blind, Placebo-controled Parallel Group Efficacy and Safety Study of BI 1356 (5 mg Administered Orally Once Daily) Over 24 Weeks, in Drug Naive or Previously Treated (6 Weeks Washout) Type 2 Diabetic Patients With Insufficient Glycemic Control
Brief Title: Efficacy and Safety of BI 1356 (Linagliptin) Versus Placebo in Type 2 Diabetic Patients With Insufficient Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.16; 2007-002448-10 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-01-14; First posted 2008-02-22 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- linagliptin 5 mg (Experimental): linagliptin 5 mg once daily
  Interventions: Drug: linagliptin
- placebo (Placebo Comparator): placebo matching linagliptin 5 mg tablets
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: linagliptin — active
  Arms: linagliptin 5 mg
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
To investigate efficacy, safety and tolerability of BI 1356 versus placebo

ELIGIBILITY:
Inclusion criteria:

* Male or female patients with type 2 diabetes and insufficient glycaemic control.
* Age 18 or over and not older than 80 years

Exclusion criteria:

* Use of more than one oral antidiabetic agent within 10 weeks prior to informed consent, insulin, glitazones or GLP-1 analogues within 3 months.
* Myocardial infarction, stroke or transient ischaemic attack within 6 months prior to informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (69):
- Croatia (2):
  - 1218.16.38605 Boehringer Ingelheim Investigational Site, Krapinske Toplice
  - 1218.16.38604 Boehringer Ingelheim Investigational Site, Slavonski Brod
- India (14):
  - 1218.16.91009 Boehringer Ingelheim Investigational Site, Andhra Pradesh
  - 1218.16.91002 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.16.91005 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.16.91014 Boehringer Ingelheim Investigational Site, Chennai
  - 1218.16.91013 Boehringer Ingelheim Investigational Site, Ghaziabad
  - 1218.16.91010 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1218.16.91006 Boehringer Ingelheim Investigational Site, Jaipur
  - 1218.16.91011 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1218.16.91008 Boehringer Ingelheim Investigational Site, Mangalore
  - 1218.16.91007 Boehringer Ingelheim Investigational Site, Manipal
  - 1218.16.91004 Boehringer Ingelheim Investigational Site, Mumbai
  - 1218.16.91003 Boehringer Ingelheim Investigational Site, Nashik
  - 1218.16.91012 Boehringer Ingelheim Investigational Site, Tamilnadu
  - 1218.16.91001 Boehringer Ingelheim Investigational Site, Trivandrum, Kerala
- Israel (6):
  - 1218.16.97267 Boehringer Ingelheim Investigational Site, Giv‘atayim
  - 1218.16.97263 Boehringer Ingelheim Investigational Site, Haifa
  - 1218.16.97265 Boehringer Ingelheim Investigational Site, Holon
  - 1218.16.97261 Boehringer Ingelheim Investigational Site, Jerusalem
  - 1218.16.97262 Boehringer Ingelheim Investigational Site, Nahariya
  - 1218.16.97266 Boehringer Ingelheim Investigational Site, Safed
- Italy (5):
  - 1218.16.39004 Boehringer Ingelheim Investigational Site, Catanzaro
  - 1218.16.39008 Boehringer Ingelheim Investigational Site, Genova
  - 1218.16.39002 Boehringer Ingelheim Investigational Site, Milan
  - 1218.16.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 1218.16.39006 Boehringer Ingelheim Investigational Site, Roma
- Malaysia (7):
  - 1218.16.60006 Boehringer Ingelheim Investigational Site, Alor Star
  - 1218.16.60003 Boehringer Ingelheim Investigational Site, Kelantan Kota Bahru
  - 1218.16.60001 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1218.16.60002 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 1218.16.60004 Boehringer Ingelheim Investigational Site, Perak
  - 1218.16.60005 Boehringer Ingelheim Investigational Site, Perak
  - 1218.16.60007 Boehringer Ingelheim Investigational Site, Pulau Pinang
- Netherlands (10):
  - 1218.16.31009 Boehringer Ingelheim Investigational Site, Andijk
  - 1218.16.31024 Boehringer Ingelheim Investigational Site, Castricum
  - 1218.16.31006 Boehringer Ingelheim Investigational Site, Deurne
  - 1218.16.31001 Boehringer Ingelheim Investigational Site, Ewijk
  - 1218.16.31010 Boehringer Ingelheim Investigational Site, Losser
  - 1218.16.31003 Boehringer Ingelheim Investigational Site, Oude Pekela
  - 1218.16.31021 Boehringer Ingelheim Investigational Site, Poortvliet
  - 1218.16.31004 Boehringer Ingelheim Investigational Site, Rijswijk
  - 1218.16.31008 Boehringer Ingelheim Investigational Site, Roelofarendsveen
  - 1218.16.31002 Boehringer Ingelheim Investigational Site, Wildervank
- Poland (3):
  - 1218.16.48603 Boehringer Ingelheim Investigational Site, Lublin
  - 1218.16.48601 Boehringer Ingelheim Investigational Site, Warsaw
  - 1218.16.48604 Boehringer Ingelheim Investigational Site, Zabrze
- Romania (2):
  - 1218.16.40604 Boehringer Ingelheim Investigational Site, Brasov
  - 1218.16.40603 Boehringer Ingelheim Investigational Site, Galati
- Slovakia (6):
  - 1218.16.42103 Boehringer Ingelheim Investigational Site, Banská Bystrica
  - 1218.16.42102 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.16.42104 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.16.42105 Boehringer Ingelheim Investigational Site, Bratislava
  - 1218.16.42101 Boehringer Ingelheim Investigational Site, Nové Mesto nad Váhom
  - 1218.16.42106 Boehringer Ingelheim Investigational Site, Šamorín
- Thailand (2):
  - 1218.16.66001 Boehringer Ingelheim Investigational Site, Bangkok
  - 1218.16.66002 Boehringer Ingelheim Investigational Site, Khon Kaen
- Ukraine (12):
  - 1218.16.38011 Boehringer Ingelheim Investigational Site, Dnipro
  - 1218.16.38002 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.16.38004 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.16.38010 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1218.16.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.16.38005 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.16.38008 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.16.38009 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.16.38012 Boehringer Ingelheim Investigational Site, Kiev
  - 1218.16.38003 Boehringer Ingelheim Investigational Site, Lviv
  - 1218.16.38006 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1218.16.38007 Boehringer Ingelheim Investigational Site, Zaporizhzhya

REFERENCES:
- [Derived] Del Prato S, Patel S, Crowe S, von Eynatten M. Efficacy and safety of linagliptin according to patient baseline characteristics: A pooled analysis of three phase 3 trials. Nutr Metab Cardiovasc Dis. 2016 Oct;26(10):886-92. doi: 10.1016/j.numecd.2016.06.015. Epub 2016 Jul 1. PMID 27484756
- [Derived] Johansen OE, Neubacher D, von Eynatten M, Patel S, Woerle HJ. Cardiovascular safety with linagliptin in patients with type 2 diabetes mellitus: a pre-specified, prospective, and adjudicated meta-analysis of a phase 3 programme. Cardiovasc Diabetol. 2012 Jan 10;11:3. doi: 10.1186/1475-2840-11-3. PMID 22234149

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients randomized to receive treatment with matching placebo
- Linagliptin: Patients randomized to receive treatment with Linagliptin 5mg
Period: Overall Study
Arm/Group | Placebo | Linagliptin
Started | 167 (number who started treatment) | 336 (number who started treatment)
Completed | 152 (number who completed treatment) | 318 (number who completed treatment)
Not Completed | 15 | 18
Not completed — Adverse Event | 4 | 5
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 4 | 6
Not completed — Other incl. lack of efficacy | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin | Total
Number analyzed (Participants) | 167 | 336 | 503
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (10.3) | 56.4 (10.1) | 55.7 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 172 | 260
  Male | 79 | 164 | 243
Body Mass Index (BMI) continuous [Mean (Standard Deviation); unit: kg/m^2] | 29.08 (4.84) | 29.04 (4.80) | 29.05 (4.81)
Glycosylated Hemoglobin A1 (HbA1C) [Mean (Standard Deviation); unit: Percent] | 8.00 (0.86) | 8.00 (0.87) | 8.00 (0.67)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 168.7 (39.3) | 164.7 (41.9) | 166.0 (41.1)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 24
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 333
Percent | 0.25 (0.07) | -0.44 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.69, 95% CI [-0.85 to -0.53], Standard Error of Mean 0.08

2. Secondary Outcome: HbA1c Change From Baseline at Week 6
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 6 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 333
Percent | 0.09 (0.05) | -0.37 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.46, 95% CI [-0.58 to -0.34], Standard Error of Mean 0.06

3. Secondary Outcome: HbA1c Change From Baseline at Week 12
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 12 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 333
Percent | 0.16 (0.06) | -0.46 (0.04)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.61, 95% CI [-0.76 to -0.47], Standard Error of Mean 0.08

4. Secondary Outcome: HbA1c Change From Baseline at Week 18
Description: HbA1c is measured as a percentage. Thus, this change from baseline reflects the Week 18 HbA1c percent minus the baseline HbA1c percent. Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 333
Percent | 0.21 (0.07) | -0.45 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -0.66, 95% CI [-0.82 to -0.49], Standard Error of Mean 0.08

5. Secondary Outcome: FPG Change From Baseline at Week 24
Description: This change from baseline reflects the Week 24 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: This population includes the FAS using the LOCF imputation, with the further restriction of patients with a baseline and post-baseline FPG value.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 149 | 318
mg/dL | 14.84 (2.98) | -8.47 (2.03)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -23.31, 95% CI [-30.37 to -16.26], Standard Error of Mean 3.59

6. Secondary Outcome: FPG Change From Baseline at Week 6
Description: This change from baseline reflects the Week 6 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 6
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 149 | 318
mg/dL | 6.73 (2.33) | -10.87 (1.59)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -17.60, 95% CI [-23.11 to -12.08], Standard Error of Mean 2.81

7. Secondary Outcome: FPG Change From Baseline at Week 12
Description: This change from baseline reflects the Week 12 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 12
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 149 | 318
mg/dL | 10.23 (2.63) | -10.75 (1.80)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -20.98, 95% CI [-27.21 to -14.75], Standard Error of Mean 3.17

8. Secondary Outcome: FPG Change From Baseline at Week 18
Description: This change from baseline reflects the Week 18 FPG minus the baseline FPG. Means are treatment adjusted for baseline HbA1c, baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and week 18
Population: as for outcome 5
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 149 | 318
mg/dL | 13.11 (2.82) | -7.25 (1.93)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -20.36, 95% CI [-27.05 to -13.68], Standard Error of Mean 3.40

9. Secondary Outcome: Percentage of Patients With HbA1c <7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7.0% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 7.0%. Only patients with baseline HbA1c >= 7%
Time Frame: Baseline and week 24
Population: This population includes the FAS with baseline HbA1c >= 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 147 | 306
percentage of patients | 11.6 (0) | 25.2 (0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 2.869, 95% CI [1.575 to 5.225]

10. Secondary Outcome: Percentage of Patients With HbA1c<7.0% at Week 24
Description: The percentage of patients with an HbA1c value below 7.0% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 7.0%.
Time Frame: Baseline and week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 333
percentage of patients | 15.3 | 28.2

11. Secondary Outcome: Percentage of Patients With HbA1c <6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 6.5%. Only patients with baseline HbA1c >= 6.5%.
Time Frame: Baseline and week 24
Population: This population includes the FAS with baseline HbA1c >= 6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 162 | 329
percentage of patients | 4.9 (0) | 10.6 (0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.0323, Regression, Logistic; Odds Ratio (OR) = 2.436, 95% CI [1.078 to 5.507]

12. Secondary Outcome: Percentage of Patients With HbA1c<6.5% at Week 24
Description: The percentage of patients with an HbA1c value below 6.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c >= 6.5%.
Time Frame: Baseline and week 24
Population: This population includes the Full Analysis Set (FAS). Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Percentage of Patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 333
Percentage of Patients | 4.9 | 10.8

13. Secondary Outcome: Percentage of Patients With HbA1c Lowering by 0.5% at Week 24
Description: The percentage of patients with an HbA1c reduction from baseline >= 0.5% at week 24 was calculated for each treatment arm. If a patient did not have an HbA1c value at week 24 they were considered a failure, so HbA1c reduction less than 0.5%.
Time Frame: Baseline and week 24
Population: The Full Analysis Set (FAS) included all patients with a baseline and at least one on treatment HbA1c measurement available. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 163 | 333
percentage of patients | 19.0 (0) | 47.1 (0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 4.243, 95% CI [2.665 to 6.755]

14. Secondary Outcome: Adjusted Means for 2h Post Prandial Blood Glucose (PPG) Change From Baseline at Week 24
Description: This change from baseline reflects the Week 24 2h PPG minus the baseline 2h PPG. Means are treatment adjusted for baseline HbA1c, baseline PPG and previous anti-diabetic medication.
Time Frame: Baseline and week 24
Population: Meal Tolerance Test (MTT) set (patients with adequate MTT results available at the beginning and end of the randomised treatment period)
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin
Number analyzed (Participants) | 24 | 67
mg/dL | 24.87 (10.33) | -33.51 (6.19)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin; Linagliptin vs. Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -58.38, 95% CI [-82.33 to -34.43], Standard Deviation 12.05

ADVERSE EVENTS:
Time Frame: From day of first drug dose until 7 days after last dose, an average of 167 days
Arm/Group | Placebo | Linagliptin
Serious Adverse Events (participants affected / at risk) | 7/167 | 10/336
Other Adverse Events (participants affected / at risk) | 38/167 | 29/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=167) | Linagliptin (N=336)
Atrial fibrillation (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Cellulitis pharyngeal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1
Platelet count decreased (Investigations) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=167) | Linagliptin (N=336)
Hyperglycaemia (Metabolism and nutrition disorders) | 38 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.